CLINICAL TRIAL: NCT04487288
Title: Added Value in Combined Use of Fusion Imaging and Contrast-enhanced Ultrasonography Compared to Fusion Imaging Alone for Percutaneous Biopsies of Focal Liver Lesions
Brief Title: Added Value in Combined Use of Fusion Imaging and Contrast-enhanced Ultrasonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Liver Cancer Association (Unknown)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2003-044-1108
Record Dates: First submitted 2020-07-20; First posted 2020-07-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Contrast Media, Liver, Biopsy, Fusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEUS with fusion (Experimental): Control group: The historic cohort is used to compare the results of the biopsy using fusion only technique from 2013 to 2019.
  Interventions: Diagnostic Test: SONAZOID

INTERVENTIONS:
Diagnostic Test: SONAZOID — CEUS using SONAZOID with fusion technique

SUMMARY:
So far, there have been studies showing that the CEUS-grafted technique has added value in biopsy and RFA, but no studies have compared the group using only fusion and the group using CEUS+fusion. Therefore, the additional added value of CEUS will be evaluated by comparing the two groups.

DETAILED DESCRIPTION:
Despite the rapid development of tumor markers and liver imaging, pathological confirmation is still necessary for atypical liver lesions that do not meet imaging criteria. US guided procedures are widely used as a method to identify focal lesions of the liver pathologically, and these US guided procedures have no burden on the operation, can be easily accessed, and have a lower cost than surgery. However, the frequency of pathological confirmation with this US guided procedure remains at around 90%. In order to increase this probability, a technique for fusion of liver CT/MRI and US has been widely used in recent years, and this allows accurate targeting of small lesions through structures seen in CT and MR. Through the fusion technique, the biopsy success rate for focal lesions can be increased to 94.4%. However, there are many cases where lesions deeply located in patients with cirrhosis are invisible, and biopsy is difficult only with fusion due to poor sonic window in patients with high BMI. To this end, a technique called contrast-enhanced ultrasonography (CEUS), such as the fusion technique, was added, which is a technique that can identify tumor vascularity in real-time using second-generation contrast media. In recent studies, there are studies combining this fusion technique and CEUS technique, and the success rate of these techniques varies from 87.6% to 97.5%. Although CEUS with fusion techniques are theoretically superior to fusion only technique, the use of CEUS adds cost of contrast media and is limited in patients with side effects on contrast media. . Also, there is no study comparing the two so far, and this study intends to compare the technique combining CEUS and fusion and the technique using only fusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ultrasound biopsy to confirm local liver lesions
* Adults over 18
* Patients who underwent multi-phasic liver CT or MRI within 6 weeks prior to the procedure
* Patients who understand and agree to the explanation and consent form and submit the consent form

Exclusion Criteria:

* Non-adaptive patients with ultrasound contrast agents (eg acute respiratory failure, heart disease, egg allergy, pregnant women, lactating women)
* Those who have difficulty obtaining proper liver ultrasound images A. Patient cooperation is not possible B. If it is difficult to obtain an image that is appropriate for the researcher's judgment (atrophy of the right lobe of the liver, a bowel is located between the liver and the abdominal wall, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Biopsy yield rate | about 2weeks
  Yield rate

SECONDARY OUTCOMES:
Complication rate | about 2days
  Complication rate
Tumor visibility on B-mode US | immediately
  Tumor visibility on B-mode US which divided into 1 (no visualization), 2 (poorly visible), 3 (indistinct), and 4 (clearly visible)
Evaluation of safety access routes to avoid complication | Time: immediately
  Evaluate whether the needle has a safety route that can prevent complication by avoiding vessels or bile ducts in the liver.
Tumor vascularity on CEUS | Time: immediately
  The tumor vascularity is evaluated by CEUS (hyper, iso, hypo vascularity on arterial phase), and compared to contrast enhancement on the CT or MRI
Subjective evaluation on the success of the procedure | immediately
  Immediately after the procedure, the reliability of appropriate tissue collection for the viable portion is determined and recorded. A score of 3-4 means that operator is expecting a successful enough tissue harvest, and a score of 1-2 means operator is not expecting proper tissue collection.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, PhD, Principal Investigator — Seoul National University Hospital, Radiology department
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No